CLINICAL TRIAL: NCT05363956
Title: Antiplaque Efficacy of Two Novel Commercially Available Herbal Toothpastes.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ajman University (Other)
Responsible Party: Principal Investigator, sudhir rama varma, Clinical Assistant Professor, Ajman University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: D-H-S-2021-NOV-24-19
Record Dates: First submitted 2022-04-26; First posted 2022-05-06 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Gingivitis; Plaque, Dental
Keywords: gingivitis; dental plaque; herbal; dentifrice; miswak; eucalyptol
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Eucalyptus Oil

STUDY DESIGN:
Intervention Model Description: The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique. The technique will be demonstrated to the patient and an image of the technique provided to the participants.
Who Masked: Participant
Masking Description: Patients were not told which dentifrice they will be given
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- miswak (Active Comparator): The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique. The technique will be demonstrated to the patient and an image of the technique provided to the participants.
  Interventions: Drug: salvadora; Drug: Eucalyptus Oil
- eucalyptus oil (Active Comparator): The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique. The technique will be demonstrated to the patient and an image of the technique provided to the participants.
  Interventions: Drug: salvadora; Drug: Eucalyptus Oil

INTERVENTIONS:
Drug: salvadora — The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique.
  Other Names: Miswak
Drug: Eucalyptus Oil — The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique.

SUMMARY:
Maintaining proper oral hygiene is essential in the prevention of oral as well as general illness. The use of herbal medicine in dentistry is growing exponentially over the years. Today, herbal medicine is considered an effective alternative to manufactured medication.

The objective of this current randomized control study is to assess the anti-plaque efficiency of Miswak (Salvadora Persica) and Eucalyptus toothpaste in the treatment of gingivitis.

Materials and Methods: This randomized experimental study enrolled 30 healthy individuals as controls and 30 individuals with mild to moderate gingivitis. The study lasted 20 days and included a two-week washout period between Miswak and Eucalyptus toothpaste. The gingival and plaque index were measured at specific time intervals during the research period.

DETAILED DESCRIPTION:
The Ajman University Ethical Committee accepted the current randomized trial; the reference number is (D-H-S-2021-NOV-24-19). The research was conducted from January 1, 2022, to March 1, 2022. The current study was carried out following CONSORT standards and the Helsinki Declaration as updated in 2013. The following kinds of toothpaste were used in this randomized crossover clinical study: Miswak toothpaste (Dabur, India) contains contains primarily miswak, with traces of other elements; Eucalyptus toothpaste (Eucalyptus-Bio (Argiletz, France)) contains primarily eucalyptus, with traces of other elements Patient Selection The PS program online version 3.16 (power and sample size calculations) was used to calculate the sample size. The inclusion criteria included subjects who are medically fit, subjects with gingival inflammation not progressed into periodontitis, and subjects between the age of 20-and 60 years. The exclusion criteria included subjects who are medically compromised, subjects on active treatment of antibiotics and corticosteroids, subjects with periodontitis (according to the AAP 2017 classification), subjects who have undergone a periodontal therapy for the past 3 months, and subjects who are healthy but have been using herbal dentifrices. A total of 120 subjects were examined However, only Thirty gingivitis patients and thirty healthy patients to be used as a control met the inclusion criteria.

Study Design This crossover randomized single-blinded study was conducted with a 20-day total examination period. The individuals were informed in great detail about the necessity for clinical evaluation for research objectives, and a signed agreement was acquired. A sample size of 30 patients with gingivitis was selected and the other 30 patients without gingivitis were used as a control. Randomization to which study group participants will belong was done by drawing lots into either the test 1 (Dabur Miswak, India), test 2(Eucalyptus-Bio, Argiletz, France), or the Active control group. To achieve blinding, serial opaque cardboard boxes with pre-assigned numbers corresponding to the Lot randomization code will be utilized to assign participants to their appropriate groups. After being assigned to their respective groups, the participants were blinded. On the first (baseline) day of the trial, all individuals were subjected to an oral examination. The baseline score was obtained for patients who met the inclusion criteria at the beginning of the study and followed up throughout the study.

The participants were given a dentifrice that had been labeled and tagged with a number. All participants were asked to brush their teeth twice daily with a 1cm line of paste in their respective brushes for two minutes, once in the morning and the other at night, using the modified bass technique. The technique will be demonstrated to the patient and an image of the technique provided to the participants. The Oral hygiene index(Plaque index) of the facial surface of three maxillary teeth, the lingual surface of the two posterior mandibular teeth, and the labial surface of one anterior mandibular tooth were calculated (OHIS, Greene & Vermillion, 1962) and the Gingival index of all teeth (Loe and Silness 1963) were recorded at the initial appointment (baseline) in the morning. All examinations were performed in the morning and by the same examiner at all recall visits, as this helps in reducing the risk of bias and quantifying the results.

Following that, subjects were instructed to use miswak toothpaste twice a day for three days. Plaque and gingival bleeding scores were evaluated again after 72 hours. The 3 days study design was developed by Marchetti et al study the 3-day plaque accumulation model to compare the efficiency of essential oil mouthwash with and without alcohol instead of kinds of toothpaste. (Marchetti, E. et al., 2011) Another study was performed by Duarte, K. et al. in 2022 and followed the 3 days plaque accumulation model to compare the efficiency of two herbal kinds of toothpaste with closely resembles our study.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit
* gingivitis patients
* subjects between 20-60 years of age

Exclusion Criteria:

* systemically compromised
* subjects who had undergone periodontal treatment in the last 6 months
* subjects using herbal dentifrice
* subjects having periodontal disease

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Gingivitis Bleeding score | 72 hours
  The Gingivitis bleeding score of the facial surface of three maxillary teeth, the lingual surface of the two posterior mandibular teeth, and the labial surface of one anterior mandibular tooth were calculated at the initial appointment (baseline) in the morning and 72 hours later. All examinations were performed in the morning and by the same examiner at all recall visits, as this helps in reducing the risk of bias and quantifying the results.

SECONDARY OUTCOMES:
Plaque score | 72 hours
  The plaque score of the facial surface of three maxillary teeth, the lingual surface of the two posterior mandibular teeth, and the labial surface of one anterior mandibular tooth were calculated at the initial appointment (baseline) in the morning and 72 hours later. All examinations were performed in the morning and by the same examiner at all recall visits, as this helps in reducing the risk of bias and quantifying the results.

CONTACTS AND LOCATIONS:
Locations (1):
- Ajman University, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared among those researchers who are interested
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be shared immediately
Access Criteria: via email